CLINICAL TRIAL: NCT04704063
Title: A Randomized, Double-Blind, Placebo-Controlled Study, to Assess the Efficacy and Safety of Tocovid Suprabio 200mg in Non-alcoholic Fatty Liver (NAFL)
Brief Title: Efficacy and Safety of Tocovid Suprabio 200mg in Non-alcoholic Fatty Liver (NAFL)
Acronym: T3-NAFL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuen Kah Hay (Other)
Collaborators: Monash University Malaysia (Other); Hovid Berhad (Industry)
Responsible Party: Sponsor-Investigator, Yuen Kah Hay, Professor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T3-NAFL-01-2019
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hepatic Steatosis; NAFLD
Keywords: Tocotrienols; Palm tocotrienol complex; NAFLD; Hepatic Steatosis; Vitamin E; Fatty Liver
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Tocotrienols; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Tocovid Suprabio 200mg
  Interventions: Drug: Tocotrienols / Vitamin E
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: Tocotrienols / Vitamin E — Palm Tocotrienols complex
  Other Names: Tocovid Suprabio
  Arms: Active
Drug: Placebo control — Placebo matching Tocovid Suprabio
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
Palm-derived tocotrienols have shown hepatoprotective effects in both animal and human studies. This study aims to investigate the effects of tocotrienols in hepatocellular lipid content using MRI. Non-alcoholic fatty liver disease (NAFLD) is a spectrum of diseases ranging from simple fatty liver (steatosis, NAFL) to non-alcoholic steatohepatitis (NASH) to cirrhosis. NASH is the accumulation of fat in liver cells accompanied with inflammation that can lead to the scarring of the liver. Prevention of liver fibrosis by early introduction of low risk interventions such as lifestyle modification, diet control and nutraceuticals may help circumvent long-term healthcare costs associated with management of chronic NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old.
2. Diagnosis of non-alcoholic fatty liver (NAFL, hepatic steatosis), using ultrasound or Fibroscan
3. Willing to provide written informed consent

Exclusion Criteria:

1. History or evidence of medical condition(s) associated with chronic liver disease other than NAFL
2. Known history or other evidence of decompensated liver disease (Child-Pugh Grade B or higher), coagulopathy, hyperbilirubinemia, hepatic encephalopathy, hypoalbuminemia, ascites, hepatic encephalopathy, and bleeding from esophageal varices are conditions consistent with decompensated liver disease.
3. Documented underlying medical conditions which may affect assessment or follow-up as listed:

   * Any malignancies
   * eGFR < 60
   * Severe dementia or psychosis
   * Requirement of long-term corticosteroid treatment for the underlying disease such as connective tissue disease
   * Uncontrolled Hemoglobinopathy or anemia
   * Uncontrolled Hyperthyroidism or Hypothyroidism
   * Hemochromatosis
   * Hepatobiliary disorders
   * Participant underwent splenectomy or suffered from splenomegaly
   * Hepatitis B or C
4. History of drug or substance abuse.
5. Estimated alcohol consumption of more than 20 g/day (1 standard drink/day) for women or more than 30 g/day (2 standard drinks/day) for men for at least 6 months prior to enrollment, binge drinking behavior or Alcohol Use and Disorders Identification Test (AUDIT) score of 7 or more
6. History of taking medications known to cause liver impairment such as systemic glucocorticoids, tetracyclines, anabolic steroids, valproic acid, or other known hepatotoxins within 3 months prior to study enrollment
7. History of major organ transplantation with an existing functional graft.
8. Present with signs of acute infection or inflammation at Screening
9. Has medical conditions or recent procedures that do not allow for magnetic resonance (MR) assessments
10. Pregnant, breast feeding, or female of childbearing potential (unless the participant is on effective contraception methods or underwent bilateral tubal ligation, bilateral oophorectomy or hysterectomy previously)
11. Participation in any other interventional trial within the previous three months. Participants enrolled in this study cannot be enrolled in another study for either research, diagnostic or treatment purposes.
12. Known history of severe allergy or immunologically mediated disease (e.g., vasculitis, cryoglobulinemia, inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis requiring more than intermittent nonsteroidal anti-inflammatory medications for management, etc.)
13. New treatment with liver-protective supplements such as S-adenosyl methionine (SAM-e), Ursodeoxycholic acid (UDCA), betain, milk thistle (silymarin), soybean phospholipids (EssentialE®), or fish oil, within 1 month prior to study enrollment.
14. Treatment with vitamin E tocopherol (at dosage more than 50mg/day) or tocotrienols within 1 month prior to enrollment.
15. Treatment using new anti-lipidemic or anti-diabetic agents within 3 months prior to study enrollment.
16. Participant having lesions with a propensity to bleed (e.g., bleeding peptic ulcers) and those having a history of hemorrhagic stroke and those with inherited bleeding disorders (e.g., hemophilia) or patients on warfarin.
17. Elevation of AST or ALT greater than five times upper limit normal (ULN), approximately 250 IU/L, or alkaline phosphatase more than two times ULN (250-300 IU/L).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Reduction of Liver Fat (VLFF) | 12 months
  Between group difference in the proportion of patients with ≥ 30% reduction of baseline of liver fat by Magnetic Resonance Imaging - Volumetric Liver Fat Fraction (MRI-VLFF)

SECONDARY OUTCOMES:
Change in liver biochemistry | 12 months
  Between group difference in mean change of liver biochemistries (ALT, AST, GGT, AP, Bilirubin)
Change in liver fat fraction | 12 months
  Between group difference in mean change (%) from Baseline to 12 months in hepatic fat fraction by MRI-VLFF
Change in serum lipid profile | 12 months
  Between group difference in mean change of serum lipid profile
Occurrence of adverse events and serious adverse events | 12 months
  Between group difference in the occurrence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Kah Hay Yuen, PhD, Study Chair — Universiti Sains Malaysia
Locations (4):
- Malaysia (4):
  - KK Bandar Baru Air Itam, Pulau Pinang, Pulau Pinang
  - KK Jalan Perak, Pulau Pinang, Pulau Pinang
  - KK Bayan Baru, Pulau Pinang, Pulau Pinang
  - Hospital Seberang Jaya (CRC), Seberang Jaya, Pulau Pinang

IPD SHARING:
Plan to Share IPD: No